CLINICAL TRIAL: NCT00453102
Title: Phase II Study of Ibritumomab Tiuxetan (Zevalin®) in Patients With Previously Untreated Marginal Zone Lymphoma
Brief Title: Yttrium Y 90 Ibritumomab Tiuxetan and Rituximab in Treating Patients With Previously Untreated Marginal Zone Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Izidore Lossos, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20060078; SCCC-2005133 (Other: University of Miami Sylvester Comprehensive Cancer Center); WIRB-20060249 (Other: Western Institutional Review Board)
Record Dates: First submitted 2007-03-27; First posted 2007-03-28 (Estimated); Results first posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-11

CONDITIONS: Marginal Zone Lymphoma
Keywords: Marginal Zone Lymphoma; Non-gastric extranodal Marginal Zone Lymphoma; Splenic Marginal Zone Lymphoma; Nodal Marginal Zone Lymphoma; Gastric Marginal Zone Lymphoma; MZL; Non-gastric extranodal MZL; Splenic MZL; Nodal MZL; Gastric MZL
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — Rituximab; ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zevalin + Rituximab (Experimental): Ibritumomab Tiuxetan (Zevalin) + Rituximab
  Interventions: Drug: Rituximab; Drug: Ibritumomab Tiuxetan

INTERVENTIONS:
Drug: Rituximab — IV Infusion of 250mg/m² of Rituximab Within 4 hours on Days 1, 7, 8, 9 0.4 millicuries (mCi)/kilogram (kg) (14.8 megabecquerels (MBq)/kilogram (kg)) for patients with normal platelet count 0.3 mCi/kg (11.1 MBq/kg) for patients with platelet count of 100,000-149,000 cells/mm³
  Other Names: Rituxan; IDEC-C2B8; Chimeric anti-CD20 monoclonal antibody
Drug: Ibritumomab Tiuxetan — IV injection of Y-90 Zevalin® over 10 minutes on Days 1, 7, 8, 9:
  0.4 mCi/kg (14.8 MBq/kg) for patients with normal platelet count 0.3 mCi/kg (11.1 MBq/kg) for patients with platelet count of 100,000-149,000 cells/mm³
  Other Names: Zevalin

SUMMARY:
Zevalin may be an effective therapy for newly diagnosed marginal zone lymphoma (MZL).

DETAILED DESCRIPTION:
This phase II study will assess the clinical response rate to Ibritumomab Tiuxetan in patients with untreated nodal, splenic and non-gastric extranodal MZL as well as in antibiotic resistant patients with mucosa-associated lymphoid tissue (MALT) gastric lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old with previously untreated, histologically confirmed Marginal Zone Lymphoma (non-gastric extranodal MZL, splenic MZL and nodal MZL) or gastric MZL that did not respond to antibiotic therapy given up to 6 months prior to enrollment, but not less than 2 months)
* Measurable and evaluable disease
* All stages are eligible
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2 (Appendix B)
* Willing and able to provide written informed consent
* Women of childbearing potential must have a negative pregnancy test at study entry and must agree to use effective contraception while on treatment and for 6 months after treatment
* Life expectancy of at least 6 months

Exclusion Criteria:

* Prior chemotherapy, radiation therapy, immunotherapy, systemic corticosteroids, or systemic biologic anticancer therapy before beginning study treatment.
* ≥ 25% lymphoma bone marrow involvement
* Platelet count < 100,000 cells/mm³
* Neutrophil count < 1,500 cells/mm³
* Known history of HIV infection
* Pregnant or lactating (pregnancy test is required for all female patients of childbearing potential)
* Woman of childbearing potential or sexually active man unwilling to use adequate contraceptive protection.
* Physical or mental condition that makes patient unable to complete specified follow-up assessments

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Izidore S. Lossos, MD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida, United States

REFERENCES:
- [Background] Lossos IS, Fabregas JC, Koru-Sengul T, Miao F, Goodman D, Serafini AN, Hosein PJ, Stefanovic A, Rosenblatt JD, Hoffman JE. Phase II study of (90)Y Ibritumomab tiuxetan (Zevalin) in patients with previously untreated marginal zone lymphoma. Leuk Lymphoma. 2015 Jun;56(6):1750-5. doi: 10.3109/10428194.2014.975801. Epub 2014 Nov 20. PMID 25315074

RESULTS

PARTICIPANT FLOW:
Groups:
- Zevalin + Rituximab: Ibritumomab Tiuxetan (Zevalin) + Rituximab
  Rituximab: IV Infusion of 250mg/m² of Rituximab Within 4 hours on Days 1, 7, 8, 9 0.4 millicuries (mCi)/kilogram (kg) (14.8 megabecquerels (MBq)/kilogram (kg)) for patients with normal platelet count 0.3 mCi/kg (11.1 MBq/kg) for patients with platelet count of 100,000-149,000 cells/mm³
  Ibritumomab Tiuxetan: IV injection of Y-90 Zevalin® over 10 minutes on Days 1, 7, 8, 9:
  0.4 mCi/kg (14.8 MBq/kg) for patients with normal platelet count 0.3 mCi/kg (11.1 MBq/kg) for patients with platelet count of 100,000-149,000 cells/mm³
Period: Overall Study
Arm/Group | Zevalin + Rituximab
Started | 18
Completed | 16
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Data reported for only 16 of 18 participants due to 2 participants withdrawing consent.
Arm/Group | Zevalin + Rituximab
Number analyzed (Participants) | 16
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [55 to 70]
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (13)
Age, Continuous [Mean (Full Range); unit: years] | 62 [37 to 84]
Sex: Female, Male [Count of Participants; unit: Participants] — Data reported for only 16 of 18 participants due to 2 participants withdrawing consent.
  Participants
    Female | 7
    Male | 9
Disease Stage [Number; unit: participants] — Number of participants grouped by extent (reach) and location of the lymphoma at Baseline: Stage I, Stage II, Stage III and Stage IV. The stage depends on both the place where the malignant tissue is located and on systemic symptoms due to the lymphoma ("B symptoms": night sweats, weight loss of >10% or fevers).The higher the stage number, the larger the extent of the lymphoma, and/or the more it has grown into nearby tissues.
  participants
    Stage I/II | 3
    Stage III/IV | 13
Extranodal disease sites [Number; unit: participants] — Number of participants grouped by the number of sites outside of the lymph nodes where lymphoma is present at baseline.
  participants
    0, 1 sites | 11
    2 or more sites | 5
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Number of participants grouped according to their Eastern Cooperative Oncology Group (ECOG) performance status or score at baseline. The ECOG score attempts to quantify patients' general well being and level of activities of daily life. The higher the score, the less healthy the patient's general well being and lower the the patient's level of the daily activity.
  participants
    0 | 14
    1 | 2
    2 | 0
Bone Marrow involvement [Number; unit: participants] — Number of participants grouped by the presence of lymphoma cells in the bone marrow at baseline.
  participants
    Yes | 0
    No | 16
Lactate dehydrogenase (LDH) Levels [Number; unit: participants] — Number of participants grouped by serum levels of LDH at baseline.
  participants
    Normal | 14
    Elevated | 2
Bulky disease (cm) [Number; unit: participants] — Number of patients grouped by the size of large tumors or lymph nodes in centimeters (cm) present at baseline.
  participants
    5 and less cm | 9
    More than 5 cm | 7
International Prognostic Index (IPI) Risk Group [Number; unit: participants] — Number of participants grouped by their prognosis with aggressive non-Hodgkin's lymphoma. One point is assigned for each of the following risk factors:
  * Age > 60 years
  * Stage III/IV disease
  * Elevated serum LDH
  * ECOG/Zubrod performance status of 2, 3, or 4
  * > 1 extranodal site
  The sum of the points allotted correlates with the following risk groups:
  * Low risk (0-1 points) - 5-year survival of 73%
  * Low-intermediate risk (2 points) - 5-year survival of 51%
  * High-intermediate risk (3 points) - 5-year survival of 43%
  * High risk (4-5 points) - 5-year survival of 26%
  participants
    Low risk | 3
    Low/intermediate risk | 9
    Intermediate/high risk | 4
    High risk | 0
Follicular Lymphoma International Prognostic Index (FLIPI) Risk Group [Number; unit: participants] — Number of participants grouped by their prognosis with follicular lymphoma. One point is assigned for each of the following factors:
  * Age > 60 years
  * Stage III or IV disease
  * > 4 lymph node groups involved
  * Serum hemoglobin < 12 g/dL
  * Elevated serum LDH
  The sum of the points allotted correlates with the following risk groups:
  * Low risk (0-1 points) - 5 and 10-year survivals of 91% and 71%, respectively
  * Intermediate risk (2 points) - 5 and 10-year survivals of 78% and 51%, respectively
  * High risk (3-5 points) - 5 and 10-year survivals of 53% and 36%, respectively
  participants
    Low risk | 7
    Intermediate risk | 7
    High risk | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Rate of Response (ORR) in Participants Receiving Protocol Therapy.
Description: The overall response rate (ORR) including complete response (CR), complete response unconfirmed (CRu), and partial response (PR) in participants receiving protocol therapy.
Time Frame: 12 weeks post-therapy
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Zevalin + Rituximab
Number analyzed (Participants) | 16
percentage of participants | 87.5 [65.6 to 97.7]

2. Secondary Outcome: Rate of Progression-Free Survival
Description: The time from the start of protocol therapy until the first documented or confirmed disease progression, or death related to study disease, whichever is earlier.
Time Frame: End of study.
Measure: Median (Full Range); unit: months
Arm/Group | Zevalin + Rituximab
Number analyzed (Participants) | 16
months | 47.6 [4.0 to 93.3]

3. Secondary Outcome: 5-Year Rate of Progression-Free Survival (5-Year PFS)
Description: Percentage of participants still alive without disease progression five years after the date of protocol therapy initiation.
Time Frame: 5 Years
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Zevalin + Rituximab
Number analyzed (Participants) | 16
percentage of participants | 40 [19.9 to 59.5]

4. Secondary Outcome: Overall Survival (OS) Rate
Description: The time from the date of initiation of study treatment until date of death from any cause for all participants.
Time Frame: End of Study
Population: Median overall survival by Kaplan-Meier method for all patients was not attained.
Measure: Number; unit: months
Arm/Group | Zevalin + Rituximab
Number analyzed (Participants) | 16
months | NA — End of study was reached with 11 participants confirmed alive.

5. Secondary Outcome: 5 Year Rate of Overall Survival (5-Year OS)
Description: Percentage of participants still alive five years after the date of protocol therapy initiation.
Time Frame: 5 Years
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Zevalin + Rituximab
Number analyzed (Participants) | 16
percentage of participants | 71.8 [46.8 to 86.5]

6. Secondary Outcome: Number of Participants With Unacceptable Toxicity.
Description: Number of participants with treatment-related (possible, probable, or definite) grade 3 or higher non-hematologic adverse events.
Time Frame: Up to 12 weeks post-therapy
Measure: Number; unit: participants
Arm/Group | Zevalin + Rituximab
Number analyzed (Participants) | 16
participants | 2

ADVERSE EVENTS:
Arm/Group | Zevalin + Rituximab
Serious Adverse Events (participants affected / at risk) | 2/16
Other Adverse Events (participants affected / at risk) | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zevalin + Rituximab (N=16)
Upper Respiratory Infection (Grade 3) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (Grade 3) (General disorders) | 1 (1)
Abdominal Pain (Grade 3) (Gastrointestinal disorders) | 1 (1)
Sepsis (Grade 5) (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zevalin + Rituximab (N=16)
Abdominal Pain (Grade 1-2) (Gastrointestinal disorders) | 3 (4)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 2 (6)
Allergic Reaction (Injury, poisoning and procedural complications) | 3 (3)
Anorexia (Gastrointestinal disorders) | 1 (1)
Anxiety (Nervous system disorders) | 1 (1)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Back Pain (Gastrointestinal disorders) | 2 (2)
Blurred vision (Eye disorders) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Bruising (Skin and subcutaneous tissue disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Creatinine increased (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 1 (1)
Depression (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Edema limbs (Blood and lymphatic system disorders) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 6 (8)
Febrile neutropenia (Infections and infestations) | 1 (1)
Fever (General disorders) | 6 (8)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2)
Headache (General disorders) | 3 (4)
Hematoma (Vascular disorders) | 1 (2)
Hemoglobin (Blood and lymphatic system disorders) | 9 (21)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (2)
Hepatic infection (Infections and infestations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (15)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Infection, Skin (cellulites) (Skin and subcutaneous tissue disorders) | 1 (1)
Infection, Upper airway NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Joint Pain (General disorders) | 3 (3)
Joint-function (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukocytes (Blood and lymphatic system disorders) | 15 (61)
Lymphopenia (Blood and lymphatic system disorders) | 8 (18)
Metabolic/Lab - Other(Specify) (Metabolism and nutrition disorders) | 6 (17)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Myalgia (General disorders) | 3 (3)
Myelodysplasia (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Neuralgia (General disorders) | 1 (1)
Neutrophils (Blood and lymphatic system disorders) | 9 (29)
Pain in extremity (General disorders) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Petechiae (Blood and lymphatic system disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 14 (29)
PTT (Blood and lymphatic system disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Rhinitis (Immune system disorders) | 2 (2)
Rigors/chills (General disorders) | 1 (1)
Sweating (General disorders) | 1 (1)
Thrombosis/embolism (vascular access) (Vascular disorders) | 1 (1)
Tooth disorder (General disorders) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Upper respiratory infection (Infections and infestations) | 4 (4)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Data reported for only 16 of 18 enrolled participants due to 2 participants withdrawing consent.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes